CLINICAL TRIAL: NCT01961193
Title: A Comparison Between Bandage Contact Lens, Punctal Plugs and Standard Measures in Preventing Corneal Injuries Related to Exposure in Patients Admitted to the General Intensive Care Unit.
Brief Title: A Comparison Between Bandage Contact Lens, Punctal Plugs and Standard Measures in Preventing Corneal Injuries
Acronym: COMLENPLSTAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, jonatan cohen, Prof.Jonathan Cohen, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7517
Record Dates: First submitted 2013-10-01; First posted 2013-10-11 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Contact Lens and Punctal Plug in Preventing Corneal Injuries
Keywords: critically ill patients; punctal plug; corneal injuries
MeSH Terms: conditions — Corneal Injuries | interventions — Contact Lenses; Punctal Plugs

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- bandage contact lens (Experimental): A bandage contact lens will be inserted by a physician from the ophthalmology department within the first 24 hours of admission of the patient to the ICU. The position of the lens will be confirmed. The lens will remain in-situ as long as the patient is considered to require artificial lubrication or until discharge from the intensive care unit.
  Interventions: Device: contact lens
- punctal plug (Experimental): A punctal plug (Painless Silicon Plugs),will be inserted into each eye. Lubricant drops will be instilled four times daily into each eye. The punctal plug will remain in- situ as long as the patient is considered to require artificial lubrication or until discharge from the intensive care unit at which time it will be removed by a physician from the ophthalmology department.
  Interventions: Device: punctal plug
- Control group (No Intervention): Hydroxyethylcellulose drops will be inserted into each eye four times a day and erythromycin ophthalmic ointment will be applied three times a day as well.

INTERVENTIONS:
Device: contact lens — A bandage contact lens will be inserted by a physician from the ophthalmology department within the first 24 hours of admission of the patient to the ICU. The position of the lens will be confirmed. The lens will remain in-situ as long as the patient is considered to require artificial lubrication or until discharge from the intensive care unit.
  Other Names: contact bandage lens
  Arms: bandage contact lens
Device: punctal plug — A punctal plug will be inserted into each eye. Lubricant drops ethylcellulose) will be instilled four times daily into each eye. The punctal plug will remain in-situ as long as the patient is considered to require artificial lubrication or until discharge from the intensive care unit at which time it will be removed by a physician from the ophthalmology department.
  Other Names: Painless Silicon Plugs
  Arms: punctal plug

SUMMARY:
Study Rationale:

The insertion of a bandage contact lens or punctal plug in a defined group of patients admitted to the ICU may be more effective than standard care in decreasing the incidence of corneal injuries.

Study Objectives:

1. To document the effect of a contact bandage lens and punctal plug in preventing corneal injuries in critically ill patients admitted to the ICU.
2. To assess the safety of a contact bandage lens and punctal plug in critically ill patients.

DETAILED DESCRIPTION:
This is a prospective, randomized study

Study Population:

Consecutive patients admitted to the General Intensive Care Unit of the Rabin Medical Center and Sharon Hospital Medical Center over a 6-month period who meet criteria for inclusion.

Procedures:

Consecutive patients meeting inclusion criteria will be enrolled in the study. Patients will be randomized to 3 groups: the bandage contact lens group, who will be assigned to insertion of a bandage contact lens; the punctal plug group, who will be assigned to the insertion of punctal plugs; and the control group, who will be assigned to standard eye care as currently practiced in the ICU.

In addition, patients in the study will be examined every 4 days by a physician from the ophthalmology department and at either discharge from the ICU or at time of death.

ELIGIBILITY:
Inclusion Criteria:

- Patients must be > 18 years of age. Patients who meet the following criteria will be considered eligible for the study: i) require mechanical ventilation; ii) require continuous infusion of sedative medication with or without neuromuscular paralysis; iii) anticipated ICU stay > 5 days.

Exclusion Criteria:

- Patients will be excluded if there is any preexisting corneal disease or an ophthalmic injury related to the present admission (e.g. ophthalmic trauma) to the ICU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of corneal damage | From date of randomization until date of dischrage from ICU or date of death from any cause whichever came first assessed up to 2 months.
  To document the effect of a contact bandage lens and punctal plug in preventing corneal injuries in critically ill patients admitted to the ICU.

SECONDARY OUTCOMES:
Presence of infection | From date of randomization until date of dischrage from ICU or date of death from any cause whichever came first assessed up to 2 months
  Results of bacterial cultures

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Cohen, MD Prof, Principal Investigator — ICU dep't , Rabin MC Campus Beilinson
Locations (1):
- Rabin MC Beilinson, Petah Tikva, Israel